CLINICAL TRIAL: NCT01363752
Title: A Multicenter, Two Arm, Randomized, Open Label Clinical Study Investigating Renal Function in an Advagraf® Based Immunosuppressive Regimen With or Without Sirolimus in Kidney Transplant Patients
Brief Title: A Study Looking at Kidney Function in Kidney Transplant Recipients Who Are Taking Anti-rejection Medication Including Tacrolimus and With or Without Sirolimus.
Acronym: ADHERE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PMR-EC-1212; 2010-019639-37 (EudraCT Number)
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplantation
Keywords: Kidney; Kidney Failure, Acute; Astagraf XL; Immunosuppression; Advagraf; Tacrolimus; Transplant
MeSH Terms: conditions — Acute Kidney Injury | interventions — Mycophenolic Acid; Sirolimus; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Advagraf + MMF + Steroids (Active Comparator): Without sirolimus
  Interventions: Drug: Advagraf; Drug: Mycophenolate Mofetil; Drug: Corticosteroids
- Advagraf + MMF + Steroids + Sirolimus (Experimental): With sirolimus; MMF withdrawn on Day 28; Sirolimus introduced on Day 28
  Interventions: Drug: Advagraf; Drug: Mycophenolate Mofetil; Drug: Sirolimus; Drug: Corticosteroids

INTERVENTIONS:
Drug: Advagraf — oral
  Other Names: FK506E; Prolonged release tacrolimus
Drug: Mycophenolate Mofetil — oral
  Other Names: CellCept
Drug: Sirolimus — oral
  Other Names: Rapamune
  Arms: Advagraf + MMF + Steroids + Sirolimus
Drug: Corticosteroids — i.v. and oral

SUMMARY:
The purpose of this study is to compare the effect of two anti-rejection therapy regimens on kidney function in kidney transplant recipients.

DETAILED DESCRIPTION:
This study will evaluate the potential to reduce nephrotoxic calcineurin inhibitors (CNI) therapy by lowering tacrolimus exposure from Advagraf® in combination with the non-nephrotoxic immunosuppressant sirolimus to avoid the risk of acute graft rejection, compared with an Advagraf® and Mycophenolate Mofetil (MMF) immunosuppressive regimen.

ELIGIBILITY:
Inclusion Criteria:

* End stage kidney disease and a suitable candidate for primary renal transplantation or re-transplantation (unless the graft was lost from rejection within 6 months)
* Receiving a kidney transplant from a deceased or living (non Human Leukocyte Antigen [HLA] identical) donor with compatible ABO blood type
* Female subject of childbearing potential has a negative serum or urine pregnancy test at enrollment
* Female and male subjects agree to maintain highly effective birth control during the study and for 90 days after discontinuation of dosing with study drugs. A highly effective method of birth control is defined as those which result in a low failure rate (CPMP/ ICH/ 286/ 95 modified) of less than 1% per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, some Intrauterine Devises (IUDs), sexual abstinence or vasectomized partner

Exclusion Criteria:

* Receiving or having previously received an organ transplant other than a kidney
* Cold ischemia time of the donor kidney > 30 hours
* Panel Reactive Antibody (PRA) >20%
* Receiving a graft from a non-heart-beating donor other than of Maastricht category 3 (withdrawal of support awaiting cardiac arrest)
* Significant liver disease, defined as having continuously elevated SGPT/ ALT and/ or SGOT/ AST and/ or total bilirubin levels ≥ 2 times the upper value of the normal range of the investigational site or is receiving a graft from a hepatitis C or B positive donor
* Requiring initial sequential or parallel therapy with immunosuppressive antibody preparation(s)
* Requiring ongoing dosing with a systemic immunosuppressive drug prior to transplantation (other than minimal levels of immunosuppression following failure of previous transplantation without nephrectomy)
* Significant, uncontrolled concomitant infections and/ or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or active peptic ulcer
* Pregnant woman or breast-feeding mother
* Subject or donor known to be HIV positive
* Known allergy or intolerance to tacrolimus, macrolide antibiotics, corticosteroids, sirolimus, MMF or any of the product excipients or iodine
* Evidence of malignant disease within the last 5 years, not including non-malignant skin cancers
* Currently participating in another clinical trial, and/ or has taken an investigational drug within 28 days prior to enrollment
* Unlikely to comply with the visits scheduled in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 853 (Actual)
Dates: Start 2011-03-08 (Actual); Primary Completion 2013-09-18 (Actual); Study Completion 2013-09-18 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (GFR) estimated by iohexol clearance at Week 52 post kidney transplantation | up to 1 year

SECONDARY OUTCOMES:
Efficacy failure | up to 1 year
  Composite endpoint defined as graft loss (re-transplantation, nephrectomy, death or dialysis ongoing at the study end) or subject withdrawal
GFR at Week 52 post kidney transplantation by Modification Diet in Renal Disease (MDRD) formula | up to 1 year
GFR at Week 52 post kidney transplantation by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula | up to 1 year
Calculated creatinine clearance at Week 52 post kidney transplantation by Cockcroft and Gault formula | up to 1 year
Incidence of clinical acute rejection | up to 1 year
Time to clinical acute rejection | up to 1 year
Incidence of Biopsy Confirmed Acute Rejection | up to 1 year
Time to Biopsy Confirmed Acute Rejection | up to 1 year
Subject survival | up to 1 year
Graft survival | up to 1 year
New Onset Diabetes Mellitus (NODM) as per American Diabetic Association (ADA) criteria | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe Ltd.
Locations (58):
- Australia (2):
  - 5042, New Lambton
  - 5043, Perth
- Austria (3):
  - 1141, Innsbruck
  - 1142, Linz
  - 1140, Vienna
- 3240, Minsk, Belarus
- Belgium (2):
  - 1241, Leuven
  - 1240, Liège
- Czechia (2):
  - Site 1441, Brno
  - 1440, Ostrava - Poruba
- France (10):
  - 1752, Amiens
  - 1740, Brest
  - 1742, Clermont-Ferrand
  - 1746, Créteil
  - 1750, Dijon
  - 1741, Le Kremilin Bicetre Cedex
  - 1749, Paris
  - 1751, Toulouse
  - 1748, Tours
  - 1745, Vandœuvre-lès-Nancy
- Germany (11):
  - 1541, Bochum
  - 1542, Erlangen
  - 1543, Essen
  - 1544, Frankfurt
  - 1545, Hannoversch Münden
  - 1540, Hanover
  - 1546, Heidelberg
  - 1547, Kiel
  - 1548, Leipzig
  - 1549, München
  - 1550, Münster
- 5441, Hong Kong, Hong Kong
- 1940, Budapest, Hungary
- Italy (3):
  - 2144, Palermo
  - 2143, Roma
  - 2140, Siena
- 2440, Maastricht, Netherlands
- Poland (3):
  - 2643, Katowice
  - 2640, Lodz
  - 2641, Poznan
- Russia (4):
  - 2841, Kemerovo
  - 2843, Moscow
  - 2842, Omsk
  - 2840, Vol'ginskiy
- South Korea (5):
  - 5245, Busan
  - 5243, Daegu
  - 5242, Seoul
  - 5241, Seoul
  - 5244, Seoul
- Spain (4):
  - 1640, Alicante
  - 1641, Barcelona
  - 1643, Santander
  - 1642, Vizcaya
- Taiwan (2):
  - 5343, Tainan
  - 5342, Taoyuan District
- Turkey (Türkiye) (3):
  - 3042, Istanbul
  - 3043, Istanbul
  - 3044, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=261